CLINICAL TRIAL: NCT04705441
Title: Self-management for People with Epilepsy and a History of Negative Health Events (SMART): Targeting Rural and Underserved People with Epilepsy
Brief Title: Self-management for People with Epilepsy
Acronym: SMART2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark A. Granner (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Mark A. Granner, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 201910824
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; Rural; Self-management
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention arm or waitlist arm for a period of 6 months. Participants receiving the intervention will participate in 8 web-based group sessions over Zoom led by a Nurse Educator and Peer Educator with epilepsy. The intervention will happen over 10-12 weeks and with virtual follow-up visits in both the intervention and the wait list groups. After month 6 follow-up visits have been completed (the primary study out evaluation), then the waitlist arm will start the SMART intervention and both the original SMART group and original waitlist group will be followed for an additional year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMART intervention (Experimental): Participants receiving the SMART intervention will participate in 8 group-format 45-60 minute sessions over 10-12 weeks. The intervention sessions are held over Zoom.
  Interventions: Behavioral: SMART 2
- Waitlist (No Intervention): Individuals randomized to WL will continue in their usual care. After they complete their 13-week and 6-month assessments, they will begin participating in the SMART program.

INTERVENTIONS:
Behavioral: SMART 2 — Participants receiving the SMART intervention will participate in 8 group-format 45-60 minute sessions (up to 10 participants per group), which will be collaboratively delivered over Zoom by a Nurse Educator and a Peer Educator with epilepsy. Telephone call-in and supplemental printed materials will be available for those who do not have internet access. The initial group session portion of SMART will be completed over 10-12 weeks. Educational components address the challenges imposed by epilepsy and comorbidity, as well as problem-identification and goal-setting, while Peer Educators and the group format address adherence, social support/social isolation, and self-efficacy. Following group sessions, participants will have 3 brief (no more than 15 minutes) monthly web-based or telephone maintenance sessions conducted by the Nurse Educator. Telephone sessions will address on-going issues of epilepsy self-management, including treatment adherence.
  Arms: SMART intervention

SUMMARY:
SMART is a program for adult individuals with sub-optimally controlled epilepsy. It involves educational and behavioral interventions intended to enhance epilepsy self-management.

The group sessions are conducted remotely over the teleconferencing application, Zoom. These sessions are held over an 8 week time period and are co-lead by a trained nurse educator and a trained peer educator. The peer educator is someone with epilepsy and a history of NHEs. Educators use a written curriculum delivered online, and the interactive sessions last 60-90 minutes. Groups are limited to about 6 -12 adult participants.

After the group sessions are done, individuals have 3 telephone maintenance sessions with the nurse educator once a month for the first 3 months after the group sessions end spaced approximately 4 weeks apart.

SMART is intended for adults with epilepsy, especially those who belong to disadvantaged sub groups such as rural populations, veterans with epilepsy and those who are underinsured. People with epilepsy who belong to disadvantaged sub-groups are more likely to have poor outcomes and often end up using expensive crisis-oriented care, and thus potentially might benefit the most from self-management programs if they can be actively engaged.

DETAILED DESCRIPTION:
In spite of advances in biological therapies, many people with epilepsy have poor outcomes including negative health events (NHEs), such as frequent seizures, accidents, and emergency department visits, and low quality of life. Risk factors for poorly controlled epilepsy include limited social supports, poor medication adherence, and comorbidities like mental illnesses. People with epilepsy who live in rural or under-served communities face additional challenges such as social isolation, limited access to care, and low levels of epilepsy awareness. The Managing Epilepsy Well (MEW) Network has been a national leader in developing, testing and disseminating evidence-based epilepsy self-management programs. One of these, Self-management for people with epilepsy and a history of negative health events (SMART), is a remotely-delivered group-format program that has been demonstrated to reduce NHEs and improve quality of life and physical and mental health functioning in individuals with epilepsy.

This 5-year prospective randomized controlled trial (RCT), written in response to Special Interest Project (SIP) 19-003 Managing Epilepsy Well (MEW) Network 2.0 Collaborating Center, will investigate the effects of the SMART program among people with epilepsy who have had recent NHEs vs. a 6-month wait-list control. Phase 1 is intended to set the stage for a successful RCT that will inform future dissemination and implementation efforts should RCT findings be positive. Qualitative evaluation of barriers and facilitators to participation in a self-management program as well as input from informed and committed local stakeholders will help develop a robust recruitment strategy and set of practices that will maximize engagement and retention. Phase 2, the RCT will be conducted in Iowa, led by a team from the University of Iowa, in Iowa City, Iowa in collaboration with local and regional epilepsy care stakeholders and partners. This new partnership will substantially strengthen representation of the U.S. "heartland"/Midwestern states in the MEW Network, increasing overall generalizability of MEW Network programs. Key foci of the study are to replicate the efficacy findings of the original SMART study and to obtain new information on how SMART is perceived among people with epilepsy, their families, clinicians and other stakeholders in rural and underserved communities. We hypothesize that at 6-month follow-up, SMART will be associated with a reduction in NHEs compared to wait-list control. We also expect that SMART will be associated with improved quality of life and functioning, and reduced depression, with improvement maintained at 18-month follow-up. An additional component of the proposed project is the continued development of the MEW database to supplement site-specific data and provide a source for secondary analyses including identification of patient-level and other factors that may identify individuals who may have difficulty engaging in and sustaining participation in evidence-based epilepsy self-management programs.

The University of Iowa will serve as the Institutional Review Board (IRB) of Record over one relying site, Case Western Reserve University (CWRU).

Phase 1 Procedure:

Phase 1 is intended to set the stage for a successful RCT that will inform future dissemination and implementation efforts should RCT findings be positive. Qualitative evaluation of barriers and facilitators to participation in a self-management program as well as input from informed and committed local stakeholders will help develop a robust recruitment strategy and set of practices that will maximize engagement and retention.

2-3 focus groups comprised of people with epilepsy and their family members from rural communities in Iowa will be convened to collect information on perceived barriers and facilitators to participation in an epilepsy self-management program. We will also conduct 2-3 focus groups comprised of rural health providers, social services agency administrators/staff or other professionals working in rural health. Focus groups will last 60-90 minutes in duration and will use a semi-structured interview guide adapted from previous studies in self-management of neurological conditions conducted by the CWRU investigators.

Building upon strong existing partnerships between members of the study team and epilepsy/neurological care partners across the states of Iowa and of Ohio, the study team will obtain input from relevant community stakeholders to develop an a priori recruitment and retention strategy intended to maximize enrollment of typically hard-to-reach individuals with epilepsy from underserved and rural communities. There will be 3 video-conference calls (using Zoom) prior to the RCT. Zoom is a cloud-based technology that offers a full spectrum of conferencing tools. Zoom allows the meeting organizer full control of the meeting such as muting all microphones and controlling attendees' presentation access. Attendees can virtually raise their hand allowing the session leader/instructor greater control over the collaborative classroom setting by ensuring thoughts and opinions are shared in turn. Zoom also includes a chat utility that can be used to communicate directly with the session leader/instructor or with other attendees. Given the additional features of Zoom, including the ability to have individual meeting links, breakout sessions, and phone conference bridges, this tool would be better suited to our needs than Skype Business.

In the first call, community advisory board (CAB) members (from both Iowa and Ohio) will review the SMART curriculum and identify potential barriers to recruitment and retention. In the 2nd meeting, CAB members will review the list of barriers and suggest solutions and strategies for reaching people with epilepsy who may not be initially help-seeking and discuss potential methods of retaining these individuals in the program once they are recruited. In the 3rd CAB meeting, the list of strategies will be finalized and the investigators will obtain input on how these strategies might be best operationalized. CAB meetings will be audio recorded and assessed qualitatively as a complement to the focus group findings.

Phase 2 Procedure:

SMART will consist of 8 group-format, 45-60 minute sessions (up to 10 participants per group), which will be collaboratively delivered by a Nurse Educator and a Peer Educator. The intervention will be delivered in a web-based format using a secure web teleconferencing system (such as Zoom) that will allow us to set up a virtual meeting room. Participants will be able to log on and interact via audio and/or video. Telephone call-in will be available for those who do not have internet access. Supplemental printed materials, providing the same information as provided on the web site, will be sent out in advance to the individuals who do not have internet access. Research staff will be available to help manage any difficulties that participants may have in accessing the sessions via web or telephone. Following the group-session series, participants will have 3 monthly telephone maintenance sessions lasting around 15 minutes. Maintenance session web/telephone calls will be made to study participants by a Nurse Educator with experience in epilepsy and/or chronic health condition management. Participants in both study arms will be followed for an additional 12 months after the completion of the primary comparative trial, for a total of 18 months.

Waitlist (WL) Control: Individuals randomized to WL at the conclusion of their baseline assessment will continue in their usual care. After they complete their 13-week and 6-month assessments, which are identical to the SMART group assessment, WL individuals will begin participating in the SMART intervention for the next 12 months.

Peer Educators: The PIs and the Nurse Educators will train up to 8 Peer Educators in two half-day sessions. The Peer Educators will be provided with a semi-structured "introduction" session to identify themselves and to get a chance to know each other a little better. The PI will then describe the study and the SMART intervention, reviewing each session individually. Each Peer Educator will receive a binder including all the materials to keep and review as convenient. In addition to going over each SMART session, the training will include self-care topics, communication skills, group leading/co-leading, and assistance with help-seeking pathways. This will involve role-play and repetition as needed depending on the materials and Peer Educator comfort/knowledge. Some of the Peer Educators from the previous SMART efficacy trial will be invited to serve as Peer Educators for this SMART trial in order to further increase overall group comfort and support among new Peer Educators. Since approximately 16-20 "waves" or "cohorts" of SMART groups (8-10 participants/group) will be conducted during the proposed study it is expected that each of the 8 Peer Educators will run at least 2 waves or cohorts, and some Peer Educators will run 3 or more waves or cohorts. The decision on which Peer Educator will lead a given cohort (with the Study Nurse Educator who will co-lead all sessions) will be made by consensus within the group de-briefing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Have received a previous diagnosis of epilepsy
* Be at least 18 years old
* Have experienced at least 1 NHE in the previous 6 months. NHEs that are obviously not related to having epilepsy, any other health condition, or related to personal activities or behavior (for example, being involved in a bus accident while one is a passenger on the bus) will not be counted as NHEs for this study.
* Be able to speak and understand English
* Be able to provide written, informed consent to study participation or have a legally authorized representative

Exclusion Criteria:

* Actively suicidal/homicidal
* Individuals with a diagnosis of dementia
* Individuals who are unable to provide written informed consent to participate in study and who do not have a legally authorized representative or individuals who are unable to participate in study procedures.
* Pregnant women
* Individuals who participated in Phase I of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Individual Change in NHEs | 6 months
  The proportion of individuals with change in their total numbers NHEs in the prior 6 months at baseline compared to week 24 of the trial. NHEs are defined as seizures, emergency department visits, hospitalizations, and self-harm attempts.
Total Reduction in NHEs | 6 months
  The reduction in NHE counts in the 6 months prior to baseline compared to week 24 of the trial. NHEs are defined as seizures, emergency department visits, hospitalizations, and self-harm attempts.

SECONDARY OUTCOMES:
Depressive Symptoms | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Patient Health Questionnaire-9 (PHQ-9) is a widely used and validated self-rated depression scale. The possible score range is 0-27. Higher scores mean more severe depressive symptom severity.
Functional health status | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Short Form-36 (SF-36) -- a multipurpose, short-form health survey that yields two psychometrically-based components: a physical component summary (PCS) and mental component summary (MCS).The possible score range is 0 to 100. The lower the score, the better the outcome.
Epilepsy control | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Epilepsy control will be assessed via self-reported seizure frequency.
Quality of Life Specific to Epilepsy as assessed by QOLIE-31 | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Quality of life will be assessed with the Quality of life in epilepsy (QOLIE-31) self-administered questionnaire which comprises 7 components including seizure worry, overall quality of life, emotional well-being, energy-fatigue, cognitive functioning, medication effect, and social function. The possible score range is from 0 to 100. A higher score indicates a better quality of life, therefore a better outcome.

OTHER OUTCOMES:
Confidence in Ability to Manage Epilepsy assessed by ESES | 6 months for the RCT sample, with an additional 12 month follow-up extension
  The Epilepsy Self-Efficacy Scale (ESES) 2000 version will be used to assess confidence in a participant's ability to manage epilepsy. The possible score range is 0 to 330. Higher scores mean a better outcome.
Social Support | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Social support will be measured with the Multidimensional Scale of Perceived Social Support (MSPSS), a 12-item scale that measures an individual's perception of social support provided by family and friends, as well as satisfaction with that support. The possible score range is from 12 to 84. Higher scores indicate higher perceived levels of social support.
Stigma for Epilepsy | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Stigma for Epilepsy will be measured using the 24-item Stigma Scale of Epilepsy (SSE), The SSE is a validated, versatile and sensitive instrument which has been used mainly in resource poor settings to study stigma in epilepsy. The possible score range is 0 to 100. Higher scores mean a higher perception of stigma with epilepsy.
Epilepsy Self-Management Competency | 6 months for the RCT sample, with an additional 12 month follow-up extension
  Epilepsy self-management competency will be measured with the Epilepsy Self-Management Scale (ESMS), a 38 item scale that assesses frequency of use of epilepsy self-management practices. The possible score range is 38-190. Higher scores indicate more frequent use of self-management strategies, meaning a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University; Mark Granner, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghearing GR, Briggs F, Cassidy K, Privitera M, Blixen C, Sajatovic M. A randomized controlled trial of self-management for people with epilepsy and a history of negative health events (SMART) targeting rural and underserved people with epilepsy: a methodologic report. Trials. 2021 Nov 20;22(1):821. doi: 10.1186/s13063-021-05762-z. PMID 34801061
- See also: The Managing Epilepsy Well Network's page for the SMART program — http://managingepilepsywell.org/smart